CLINICAL TRIAL: NCT04664517
Title: Casting Versus Flexible Intramedullary Nailing in Displaced Forearm Shaft Fractures in 7 to 12 Years Old Children: A Study Protocol for a Randomized Controlled Trial
Brief Title: Casting Versus Flexible Intramedullary Nailing in Displaced Pediatric Forearm Shaft Fractures
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Petra Grahn, Hand Surgeon, Principal investigator, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 78/1801/2020
Record Dates: First submitted 2020-12-06; First posted 2020-12-11 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Both Bone Forearm Fracture; AO Classification 22D/2.1-5.2; 7-12 Year Old

STUDY DESIGN:
Intervention Model Description: multicenter, randomized superiority trial. Parallell patient choice arm.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- FIN (Flexible intramedullary nail) (Active Comparator): Fracture reduction and fixation using flexible intramedullary nails. Nails size is 0.4 times the smallest diameter of the medullary canal of radius or ulna measured in radiographs.
  Interventions: Procedure: Flexible intramedullary nail (FIN)
- Long arm cast (Active Comparator): Fractures are reduced under general anesthesia within 3 days from injury and a synthetic circular above elbow cast in neutral pro-supination is applied for six weeks.
  Interventions: Procedure: Reduction auder general anesthesia and long arm cast
- Patient Choice FIN (Other): Fracture reduction and fixation using flexible intramedullary nails. Nails size is 0.4 times the smallest diameter of the medullary canal of radius or ulna measured in radiographs.
  Interventions: Procedure: Flexible intramedullary nail (FIN)
- Patient Choice cast (Other): Fractures are reduced under general anesthesia within 3 days from injury and a synthetic circular above elbow cast in neutral pro-supination is applied for six weeks.
  Interventions: Procedure: Reduction auder general anesthesia and long arm cast

INTERVENTIONS:
Procedure: Flexible intramedullary nail (FIN) — Both bone FIN
  Arms: FIN (Flexible intramedullary nail); Patient Choice FIN
Procedure: Reduction auder general anesthesia and long arm cast — Reduction and cast
  Arms: Long arm cast; Patient Choice cast

SUMMARY:
The forearm is the most common fracture location in children, with an increasing incidence. Displaced forearm shaft fractures have traditionally been treated with closed reduction and cast immobilization. Diaphyseal fractures in children have poor remodeling capacity, and malunion can thus cause permanent cosmetic and functional disability. Internal fixation especially with flexible intramedullary nails has gained increasing popularity, without evidence of a better outcome compared to closed reduction and cast immobilization.

DETAILED DESCRIPTION:
This is a multicenter, randomized superiority trial comparing closed reduction and cast immobilization to flexible intramedullary nails in 7-12 year old children with > 10° of angulation and/or > 10mm of shortening in displaced both bone forearm shaft fractures (AO-pediatric classification: 22D/2.1-5.2). A total of 78 patients with minimum 2 years of expected growth left are randomized in 1:1 ratio to either treatment group. The study has a parallel non-randomized patient preference arm. Both treatments are performed under general anesthesia. In the cast group a long arm cast is applied for 6 weeks. The flexible intramedullary nail group is immobilized in a collar and cuff sling for 4 weeks. Data is collected at baseline and at each follow-up until 1 year.

Primary outcome is 1) PROMIS Pediatric Item Bank v2.0 - Upper Extremity and 2) forearm pronation-supination range of motion at one-year follow-up. Secondary outcomes are Quick DASH, Pediatric pain questionnaire, Cosmetic VAS, wrist range of motion as well as any complications (malunion, delayed union, non-union or deep wound infection, peripheral nerve injury, need for re-intervention during 1-year follow-up) and costs of treatment.

The investigators hypothesize that flexible intramedullary nailing results in a superior outcome.

ELIGIBILITY:
Inclusion Criteria:

* 7 to12 year old children
* Open distal radial physis
* Both bone forearm shaft fractures (AO-pediatric classification: 22D/2.1-5.2)
* More than 10 degrees of angulation
* with or without less than 10mm of shortening

Exclusion Criteria:

* Patients with bilateral fractures
* Gustilo-Anderson grade I-III open fracture
* Neurovascular deficit
* Compartment syndrome
* Pathologic fracture
* Patient not able to give a written informed consent

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
PROMIS Pediatric Item Bank v2.0 - Upper Extremity | 12 months
  We aim to confirm that 75 percent of FIN patients have a better PROMIS UE score than what the mean score of the cast patients will be assuming both groups have the same standard deviation.
  PROMIS (Patient-Reported Outcomes Measurement Information System) scores are normalized to a mean score of 50, standard deviation of 10, with a theoretical range of 0 to 100. A higher score corresponds to a greater amount of the domain being measured.
Pro-supination | 12 months
  Difference (percent) in forearm pronation-supination range of motion (ROM) at one-year follow-up in comparison to uninjured side.

SECONDARY OUTCOMES:
Quick Disabilities of the Arm, Shoulder and Hand score | 6 weeks, 3, 6 and 12 months
  Minimum value is 0 and maximum 100. Higher value indicates worse function. Statistically significant difference in QuickDASH score is 6.8 (18) at 12 months FU.
Measurement Model for the Pediatric Quality of Life Inventory (PedsQL) | 6 weeks, 3, 6 and 12 months
  Minimum value is 0 and maximum value is 100. Higher score indicates better health related quality of life.
Measurement Model for the Pediatric Quality of Life Inventory Pediatric Pain Questionaire (PEDS QL PPQ) | 6 weeks, 3, 6 and 12 months
  Minimum value 0 maximum value 10. Higher value indicates higher pain intensity
Need for re-interventions | 6 weeks, 3, 6 and 12 months
  Minimum value 0 no maximum value. Lower value indicates better outcome.
Rate of participants with malunion | 6 weeks, 3, 6 and 12 months
  malunion, delayed union (defined as nonunion at 3 months or later), pseudoarthrosis (defined as 3 cortices out of 4 not united at 6 months or later)
Adverse effects | 6 weeks, 3, 6 and 12 months
  adverse effects (wound infection, nerve or/and tendon damage)
Cosmetic VAS | 6 weeks, 3, 6 and 12 months
  Minimum value 0 maximum value 10. Higher value indicates better satisfaction
PROMIS Pediatric Item Bank v2.0 - Upper Extremity | 6 weeks, 3, 6 months
  Difference between treatment groups
Upper limb ROM | 6 weeks, 3, 6 months
  Difference (percent) in elbow, wrist flexion extension and pronation-supination in comparison to uninjured side
Return to sport/musical instrument and level | 6 weeks, 3, 6 and 12 months
  Level of practiced sport or musical instrument before and at end of trial, as well as time from injury to return to hobby is registered.

CONTACTS AND LOCATIONS:
Overall Officials: Ilkka Helenius, MD, Study Director — Helsinki University Central Hospital; Petra Grahn, MD, Principal Investigator — Helsinki University Central Hospital
Locations (5):
- Finland (5):
  - HUS New Childrens Hospital, Helsinki
  - Kuopio University Hospital, Kuopio
  - Oulu University Hospital, Oulu
  - Tampere University Hospital, Tampere
  - Turku University Hospital, Turku

IPD SHARING:
Plan to Share IPD: Yes
All data will be available upon request. Data will be delivered as anonymized.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Study protocol is published in BMJ open. What can not be found there can be shared by contacting the main investigator.
Access Criteria: Please see the study protocol in BMJ open

REFERENCES:
- [Derived] Grahn P, Sinikumpu JJ, Nietosvaara Y, Syvanen J, Salonen A, Ahonen M, Helenius I. Casting versus flexible intramedullary nailing in displaced forearm shaft fractures in children aged 7-12 years: a study protocol for a randomised controlled trial. BMJ Open. 2021 Aug 20;11(8):e048248. doi: 10.1136/bmjopen-2020-048248. PMID 34417215
- See also: Protocol publication — https://bmjopen.bmj.com/